CLINICAL TRIAL: NCT06310759
Title: Observational Prospective Multicenter Validation Study Investigating the Possibility of Replacing Cystoscopies With High Volume Urine DNA Testing in Individuals With Suspicion of Urothelial Cancer (UROSCOUT-1)
Brief Title: Prospective Validation Study of High Volume Urine DNA Testing in Individuals With Suspicion of Urothelial Cancer
Acronym: UROSCOUT-1
Status: Recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other)
Responsible Party: Sponsor
Other Study IDs: R21088B
Record Dates: First submitted 2024-02-05; First posted 2024-03-15 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial neoplasms; Bladder neoplasms; Upper tract urothelial neoplasms; Liquid biopsies; Urine tumor DNA
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Urothelial cancers of the bladder and upper urinary tract account for over 200,000 deaths and 600,000 diagnoses annually worldwide. The most common presenting symptom is hematuria (blood in urine), triggering a cascade of tests, including an invasive examination of the bladder using a flexible scope (cystoscopy). Millions of cystoscopies are performed every year worldwide for patients presenting with hematuria, but only 10% result in a cancer diagnosis. The UROSCOUT-1 trial is a prospective multicenter observational study that explores the potential of urine tumor DNA (utDNA) testing to replace a significant portion of cystoscopies in the diagnostic setting for hematuria or other reasons to rule out urothelial cancer. The goal is to enhance patient quality of life, reduce healthcare costs, and address increased workloads in urology centers. Sample collection will be conducted by mail, and the samples will be analyzed in a blinded manner, without knowledge of which patients are diagnosed with cancer. Random subsampling will be applied to cancer-negative patients to achieve an approximate 1:1 ratio between cancer-positive and -negative patients.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Patient has been scheduled for cystoscopy to rule out urothelial cancer

Exclusion Criteria:

* Prior diagnosis of urothelial cancer (i.e. bladder cancer or upper tract urothelial carcinoma)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for diagnostic cystoscopy to rule out urothelial cancer due to hematuria, imaging, or urine cytology findings.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of urine tumor DNA (utDNA) test for urothelial cancer detection | 1 year after diagnostic workup
  Sensitivity and specificity of utDNA test for urothelial cancer detection, using histologically confirmed cancer diagnoses within 1 year of the diagnostic workup as ground truth

SECONDARY OUTCOMES:
Sensitivity and specificity of cystoscopy for urothelial cancer detection | 1 year after diagnostic workup
  Sensitivity and specificity of cystoscopy for urothelial cancer detection, using histologically confirmed cancer diagnoses within 1 year of the diagnostic workup as ground truth
Sensitivity and specificity of urine cytology for urothelial cancer detection | 1 year after diagnostic workup
  Sensitivity and specificity or urine cytology for urothelial cancer detection, using histologically confirmed cancer diagnoses within 1 year of the diagnostic workup as ground truth
Time to diagnosis of urothelial cancer in patients with a positive utDNA test but negative cystoscopy | 2, 5, and 10 years after diagnostic utDNA testing
  Time to diagnosis of urothelial cancer in patients with a positive utDNA test but negative cystoscopy
Adverse event rate for cystoscopy | 4 weeks after cystoscopy
  Adverse event rate for cystoscopy, based on CTCAE 5.0
Technical success rate of utDNA test | Immediately after utDNA sample analysis
  Fraction of all analyzed urine samples for which the analysis met the quality control criteria for a technically successful analysis
Estimate of diagnostic cystoscopies avoided | 4 weeks after cystoscopy
  Estimated fraction of diagnostic cystoscopies that could have been avoided by pre-screening patients with a utDNA test (calculated as the fraction of all diagnostic utDNA samples that were negative and for which subsequent cystoscopy did not lead to clinical interventions)
Specificity of high-stringency utDNA threshold | 1 year after diagnostic workup
  Specificity of a high-stringency utDNA threshold (at least 2 known urothelial cancer driver mutations with allele fraction > 5%) for clinically detectable urothelial cancer

OTHER OUTCOMES:
Characteristics of urothelial cancers that were not detected by the utDNA test | Immediately after pathological examination of surgical tissue
  Characteristics of urothelial cancers that were not detected by the utDNA test (TNM pathological stage, World Health Organization (WHO) 2004/2016 grade, and tumor size)
Concordance between utDNA and urine cytology results | Immediately after completion of utDNA analysis and urine cytology
  Concordance between utDNA and urine cytology results, with respect to positivity of the test

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Nikkola, Principal Investigator — Tampere University Hospital
Locations (8):
- Jesse Brown Department Of Veterans Affairs Medical Center, Chicago, Illinois, United States
- Vancouver Prostate Centre, Vancouver, British Columbia, Canada
- Finland (5):
  - Helsinki University Hospital, Helsinki
  - Satasairaala Hospital, Pori
  - Seinäjoki Central Hospital, Seinäjoki
  - Tampere University Hospital and Tampere University, Tampere
  - Turku University Hospital, Turku
- Kindai University Hospital, Osaka, Japan